CLINICAL TRIAL: NCT03926364
Title: Spatiotemporal Profile of Pain and Unpleasant Sensations in Referred Pain: a Feasibility Study
Brief Title: Profile of Pain and Unpleasant Sensations in Patients With Referred Pain
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Shellie A. Boudreau, Associate Professor, Aalborg University
Other Study IDs: 2015-57-0001/2
Record Dates: First submitted 2018-06-07; First posted 2019-04-24 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Referred Pain; Somatic Pain; Neuropathic Pain
Keywords: Pain drawings; referred pain; somatic pain; neuropathic pain; e-health; pain location; biopsychosocial factors; back pain; neck pain; pain extent; function
MeSH Terms: conditions — Pain, Referred; Nociceptive Pain; Neuralgia; Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Referred pain
  Interventions: Other: Patients with referred pain

INTERVENTIONS:
Other: Patients with referred pain — The project does not affect treatment or does not offer any intervention.

SUMMARY:
This feasibility study primarily aimed to assess the technology acceptance and usability of a pain tracking software in patients with spinally referred chronic pain. The secondary aim was to assess the fluctuations in pain intensity and distribution, using the pain tracking software during a 3-month period. Additionally, the study aimed to explore the patients' behavior when self-reporting pain when given the opportunity to use a variety of pain quality descriptors, such as tingling, burning and stabbing.

Patients with spinally referred chronic pain will be recruited to participate. Participants will be asked to use a pain tracking software to create weekly pain reports for a 3-month period. These pain reports consist of pain drawings and intensity scales. Additionally, patients will complete baseline disability and pain catastrophizing online questionnaires. The project does not affect treatment or does not offer any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Suffer from pain in the neck or lumbar spine referring to a limb for a more than 7 consecutive days
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Pregnancy or breastfeeding, severe infections, cancer.
* Epilepsy, Multiple sclerosis, history of stroke, diabetes, traumatic spinal cord injury resulting in permanent functions loss
* Lack of ability to cooperate due to language barrier, cognition or inability to use technology.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with referred pain recruited from advertisement in public areas, social media, public and collaborating private clinics and hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in pain extent for 3 months | 3 months
  Changes in pain extent as measured by the number of pixels drawn in digital pain drawings, at weekly intervals.

SECONDARY OUTCOMES:
Change in pain intensity for 3 months | 3 months
  Changes in usual and current pain intensity as measured by a Numerical Rating Scale, at a weekly interval.
Changes in pain location for 3 months | 3 months
  Changes of the location of pain measured by appearance and disappearance of pain in different body regions.
Disability levels at baseline | Baseline
  Description of disability levels as assessed by the Oswestry (if pain located in back) or the Neck Disability Index (if pain located in neck) online questionnaires.
Pain Catastrophizing score | Baseline
  Scores obtained from an online Pain Catastrophizing Scale (PCS) at baseline

OTHER OUTCOMES:
Demographic information | At baseline
  Online demographic information

CONTACTS AND LOCATIONS:
Overall Officials: Shellie A Boudreau, PhD, Principal Investigator — Associate Professor
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Aalborg University, Aalborg

IPD SHARING:
Plan to Share IPD: Undecided
The location of the advanced analyses may occur in collaboration with other machine learning experts